CLINICAL TRIAL: NCT04359407
Title: The Effect of Prone Positioning on Lung Aeration and Ventilation-perfusion Matching in Mechanically Ventilated Patients With Coronavirus Disease Related Acute Respiratory Distress Syndrome
Brief Title: Prone Positioning and Regional Ventilation in Mechanically Ventilated COVID-19 Patients
Acronym: COVID-19_EIT
Status: Completed | Type: Observational
Sponsor: Walid HABRE (Other)
Responsible Party: Sponsor-Investigator, Walid HABRE, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2020-00896
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; Electric Impedance; Prone Positioning
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prone positioning — Change the positioning of the COVID patients who are intubated and mechanically ventilated from supine to prone

SUMMARY:
The consensus therapeutic strategy implies that COVID patients with acute lung injury due to coronavirus are routinely placed in prone position in an attempt to improve oxygenation by increasing ventilation homogeneity. The purpose of the study is to quantify with the electrical impedance tomography (EIT) the changes in the ventilation and aeration in the dorsal regions of the lung when the patient is placed in prone position.

DETAILED DESCRIPTION:
Patients with acute respiratory distress syndrome (ARDS) frequently develop atelectasis in dorsal lung regions because of gravity and the compression by the heart and the diaphragm. Since lung perfusion is predominantly distributed in lower lung regions, a reduction of ventilation in these areas results in further ventilation-perfusion mismatch, called shunt. The development of atelectatic lung regions necessitate the use of higher ventilation pressures, which in turn results in excessive transpulmonary pressures and ventilation-induced lung injury in the ventral regions. Therefore it is common to promote the prone position in patients with ARDS in order to improve ventilation-perfusion matching and thus, protect the ventral regions from hyperinflation. In patients with COVID-19-related ARDS, the value of such therapeutic strategy based on placing in prone position has not been completely elucidated. The aims of the study are to determine whether prone positioning improves dorsal regional ventilation when compared to supine position. Moreover, another aim is to assess the changes in intrapulmonary shunt following patient position changes.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all the following criteria are eligible for the study:

* Mechanically ventilated
* Fit the Berlin Definition for moderate or severe acute respiratory distress syndrome (arterial oxygen partial pressure over inspiratory fraction of oxygen less than 200 mmHg)
* Infection with coronavirus confirmed
* Scheduled to undergo prone positioning

Exclusion Criteria:

* Patients with pacemakers, defibrillators or other electrically active implants
* Patients with damaged skin or impaired skin contact of the electrodes due to wound dressings
* Patients with chest tubes
* History of thoracic surgery or lung resection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe acute lung injury induced by the coronavirus necessitating intubation and ventilation with positioning on the ventral side.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Tidal electrical Impedance | One hour before turning to prone or supine positioning
  Change in the ratio of tidal electrical impedance variation in the dorsal and total lung areas

SECONDARY OUTCOMES:
Intrapulmonary shunt | One hour before turning to prone or supine positioning
  Changes in intrapulmonary shunt fraction
Volumetric capnography | One hour before turning to prone or supine positioning
  Changes in the phase three slope of the volumetric capnogram

CONTACTS AND LOCATIONS:
Overall Officials: Walid Habre, MD, PhD, Principal Investigator — University of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dos Santos Rocha A, Diaper J, Balogh AL, Marti C, Grosgurin O, Habre W, Petak F, Sudy R. Effect of body position on the redistribution of regional lung aeration during invasive and non-invasive ventilation of COVID-19 patients. Sci Rep. 2022 Jun 30;12(1):11085. doi: 10.1038/s41598-022-15122-9. PMID 35773299